CLINICAL TRIAL: NCT01106443
Title: Central Compartment Neck Dissection Total Thyroidectomy: a Randomized Controlled Trial
Brief Title: Central Compartment Neck Dissection With Thyroidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Peter Dziegielewski, MD, FRCSC, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88888
Record Dates: First submitted 2010-04-14; First posted 2010-04-19 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Indeterminate Thyroid Nodules
Keywords: Indeterminate thyroid nodule; fine needle aspirate biopsy; thyroidectomy; central lymph node dissection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Total Thyroidectomy - CLND (Active Comparator): Total thyroidectomy without central lymph node dissection.
  Interventions: Procedure: Total thyroidectomy - CLND
- Total Thyroidectomy +CLND (Experimental): Total thyroidectomy with central lymph node dissection.
  Interventions: Procedure: Total Thyroidectomy + CLND
- Hemi-thyroidectomy + CLND (Experimental): Hemi-thyroidectomy with central lymph node dissection.
  Interventions: Procedure: Hemi-thyroidectomy + CLND
- Hemi-thyroidectomy - CLND (Active Comparator): Hemi-thyroidectomy without central lymph node dissection.
  Interventions: Procedure: Hemi-thyroidectomy - CLND

INTERVENTIONS:
Procedure: Total Thyroidectomy + CLND — Total thyroidectomy includes removing all possible thyroid tissue. Central lymph node dissection is a neck level 6 dissection. This includes removal of all central lymphatics from carotid artery to carotid artery and hyoid to sternum/clavicle.
  Arms: Total Thyroidectomy +CLND
Procedure: Total thyroidectomy - CLND — Removal of all possible thyroid tissue without dissection of neck level 6.
  Arms: Total Thyroidectomy - CLND
Procedure: Hemi-thyroidectomy + CLND — Removal of one thyroid lobe and ipsilateral central lymph nodes
  Arms: Hemi-thyroidectomy + CLND
Procedure: Hemi-thyroidectomy - CLND — Removal of one thyroid lobe only. No lymphatic dissection.
  Arms: Hemi-thyroidectomy - CLND

SUMMARY:
When a patient presents with a thyroid mass, part of the work-up may include a fine needle aspiration biopsy (FNAB). The results of the biopsy then help plan treatment. If the results are benign, the management will typically be to follow the nodule. If the results demonstrate or are suspicious for cancer, such as papillary thyroid carcinoma (PTC), the treatment is a total thyroidectomy (total thyroid removal). The latest American thyroid association guidelines for PTC (2009) suggest that in many instances a central lymph node dissection (CLND) should be performed in conjunction with the total thyroidectomy. This procedure consists of removing the lymphatic (glandular) tissues surrounding the thyroid itself, as this tissue may have a propensity for cancer spread. The procedure's necessity has met much controversy in the last decade, but is becoming more of a standard in thyroid cancer surgery.

When a thyroid nodule FNAB is reported as indeterminate, the treatment strategy is less clear cut. While a diagnostic hemi-thyroidectomy or therapeutic total thyroidectomy may be in order, the inclusion of CLND is not clearly defined. In many centers a CLND will be omitted with surgical management for an "indeterminate" lesion, while in others, it is standard protocol. The argument of performing CLND is largely based on the tenet that it adds little surgical time, cost or risks to the patient. Because the evidence of the prognostic role of lymph node metastases is limited many would argue that the risk of not performing CLND is greater than performing CLND. Furthermore, in the event of finding cancer on final pathology, and thus, having to re-operate in the thyroid/central compartment bed, post-operative complications may increase. Opponents of CLND argue that there is a paucity of strong evidence supporting CLND in the improvement of oncologic outcomes and can potentially increase post-operative low calcium levels or vocal nerve damage However, these recommendations are based on retrospective level III evidence. Thus the debate continues: is CLND justified as an adjunct to hemi-or total thyroidectomy in indeterminate thyroid pathology?

The hypothesis is: CLND in hem- or total thyroidectomy for "indeterminate" thyroid nodules will not increase post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Indeterminate or benign pathology on fine needle aspirate biopsy
* Scheduled to undergo total or hemi-thyroidectomy
* > 18 years old

Exclusion Criteria:

* Previous thyroid surgery
* Previous neck surgery in field of thyroidectomy
* Previous neck irradiation
* Pre-operative hypocalcemia or hypoparathyroidism
* Biopsy suggestive of thyroid cancer
* Neck nodes suspicious for or with known cancer
* Pre-operative vocal cord dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Short Term Hypo-calcemia | < 1 month post-operatively
  Definition: Serum Ionized Calcium (ICa) < 0.9 mmol/L or symptoms related to hypocalcemia (acral or peri-oral paresthesia/numbness, tetany, muscle cramps/twitching, delirium etc.) and ICa < 1.0 mmol/L

SECONDARY OUTCOMES:
Long Term Hypocalcemia | > 1month
  Definition: Serum Ionized Calcium (ICa) < 0.9 mmol/L or symptoms related to hypocalcemia (acral or peri-oral paresthesia/numbness, tetany, muscle cramps/twitching, delirium etc.) and ICa < 1.0 mmol/L
Vocal Cord Dysfunction | 1 month post-operatively
  A surrogate for recurrent laryngeal nerve function. Determined pre- and post-operatively via flexible naso-pharyngoscopy (standard of care).
  - evaluated by a validated measure (Voice Handicap Index)
Positive Nodes | At the time of operation. (Time 0)
  Presence of disease with in central lymph node dissection as per pathology report.
Surgical Time | During the operation. (Time 0)
  Time from cutting skin to putting on last steri-strip on closed incision in the operating theatre.
Length of Hospital Stay | 1 day post-operatively on average
  Days spent in the hospital post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Dziegielewski, MD, Study Director — University of Alberta; Jeffrey R Harris, MD, FRCSC, Principal Investigator — University of Alberta; Robert Hart, MD, FRCSC, Study Chair — Dalhousie University; Elaine Fung, MD, Study Chair — Dalhousie University
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Dalhouise University, Halifax, Nova Scotia